CLINICAL TRIAL: NCT00097578
Title: An Observational Study of Avastin (Bevacizumab) in Combination With Chemotherapy for Treatment of Metastatic or Locally Advanced and Unresectable Colorectal Adenocarcinoma
Brief Title: A Study of Avastin With Chemotherapy for Treatment of Metastatic or Advanced and Unresectable Colorectal Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AVF2941n
Record Dates: First submitted 2004-11-24; First posted 2004-11-25 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2013-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This is an observational study designed to follow patients with metastatic or locally advanced and unresectable colorectal cancer who are receiving Avastin in combination with chemotherapy and whose cancer has been either previously untreated or treated <=4 months prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent and Authorization document
* Metastatic, or locally advanced and unresectable, adenocarcinoma of the colon or rectum
* Receiving Avastin as a component of first-line chemotherapy
* First-line chemotherapy plus Avastin initiated <=4 months prior to enrollment in the study

Exclusion Criteria:

* Patients who have contraindications for treatment with Avastin (see the Avastin Package Insert) or who would incur excessive risks with Avastin treatment are ineligible for this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Sites were selected primarily from community-based oncology practices geographically distributed across the United States.
Sampling Method: Non-Probability Sample
Enrollment: 1953 (Actual)
Dates: Start 2004-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hedrick, M.D., Study Director — Genentech, Inc.
Locations (1):
- Genentech Central Contact, South San Francisco, California, United States

REFERENCES:
- [Derived] Kabbinavar FF, Flynn PJ, Kozloff M, Ashby MA, Sing A, Barr CE, Grothey A. Gastrointestinal perforation associated with bevacizumab use in metastatic colorectal cancer: results from a large treatment observational cohort study. Eur J Cancer. 2012 May;48(8):1126-32. doi: 10.1016/j.ejca.2012.02.052. Epub 2012 Mar 15. PMID 22424880